CLINICAL TRIAL: NCT01145599
Title: Identifying Progression of Retinal Disease in Eyes With Non Proliferative Diabetic Retinopathy in Diabetes Type 2 Using Non-invasive Procedures
Brief Title: Identifying Progression of Retinal Disease in Eyes With NPDR in Diabetes Type 2 Using Non-invasive Procedures
Status: Completed | Type: Observational
Sponsor: European Vision Institute Clinical Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: ECR-RET-2010-02
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes; Non Proliferative Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type-2 diabetes, NPDR: Type-2 diabetic patients with NPDR.

SUMMARY:
The purpose of this study is to identify eyes that show worsening and disease progression (progressor phenotypes).

DETAILED DESCRIPTION:
To identify "progressors" in retinal vascular disease and central retinal edema in type 2 diabetic patients with early NPDR, based on retinal disease progression from baseline to the 12-month visit, assessed by the following biomarkers:

* Microaneurysms turnover (MA formation rate over or equal to 2, i.e. number of new MA from baseline to the 12-month visit) computed from color fundus photographs using the RetmarkerDR software; and
* Retinal thickness increase in eyes with retinal thickening (Increase in retinal thickness above normal range) in the central subfield, the inner ring and/or the outer ring Constantly Present, Present or Absent (as measured by OCT and considering the macula thickness normative data.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes type 2 according to 1985 WHO criteria
2. Age between 35 and 75 years
3. Mild non-proliferative diabetic retinopathy (levels 20 or 35, based on the ETDRS criteria) - 7 fields color fundus photography
4. Presence of at least 1 microaneurysm in the central 3000 micr. in diameter area (corresponding to 2 DA) - Field 2
5. Best Corrected Visual Acuity >= 75 letters (>= 20 /32)
6. Refraction with a spherical equivalent less than 5 Dp
7. Informed consent

Exclusion Criteria:

1. Cataract or other eye disease that may interfere with fundus examinations
2. Glaucoma
3. Any eye surgery within a period of 6-months
4. Other retinal vascular disease
5. Previous laser therapy
6. Dilatation of the pupil < 5 mm

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type-2 diabetes, NPDR
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Identify "progressors" | 12 months
  To identify "progressors" in retinal vascular disease and central retinal edema, the following 2 biomarkers will be considered: the MA formation rate (biomarker for the progression of retinal vascular disease) and the presence of retinal thickening in the central subfield and/or the inner ring (biomarker for the presence of retinal edema).

SECONDARY OUTCOMES:
Identify correlations between "progressors" and study outcomes. | 12 months
  To identify correlations between "progressors" and the different study outcomes.
  To explore the parameters, and to identify highly predictive outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: José Cunha-Vaz, MD PhD, Study Chair — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- Centre for Clinical Trials- AIBILI - Association for Innovation and Biomedical Research on Light and Image, Coimbra, Coimbra District, Portugal

REFERENCES:
- [Derived] Cunha-Vaz J, Ribeiro L, Costa M, Simo R. Diabetic Retinopathy Phenotypes of Progression to Macular Edema: Pooled Analysis From Independent Longitudinal Studies of up to 2 Years' Duration. Invest Ophthalmol Vis Sci. 2017 May 1;58(6):BIO206-BIO210. doi: 10.1167/iovs.17-21780. PMID 28785768
- [Derived] Cunha-Vaz J, Santos T, Ribeiro L, Alves D, Marques I, Goldberg M. OCT-Leakage: A New Method to Identify and Locate Abnormal Fluid Accumulation in Diabetic Retinal Edema. Invest Ophthalmol Vis Sci. 2016 Dec 1;57(15):6776-6783. doi: 10.1167/iovs.16-19999. PMID 27978559
- [Derived] Ribeiro L, Bandello F, Tejerina AN, Vujosevic S, Varano M, Egan C, Sivaprasad S, Menon G, Massin P, Verbraak FD, Lund-Andersen H, Martinez JP, Jurgens I, Smets E, Coriat C, Wiedemann P, Agoas V, Querques G, Holz FG, Nunes S, Neves C, Cunha-Vaz J; Evicr Net Study Group. Characterization of Retinal Disease Progression in a 1-Year Longitudinal Study of Eyes With Mild Nonproliferative Retinopathy in Diabetes Type 2. Invest Ophthalmol Vis Sci. 2015 Aug;56(9):5698-705. doi: 10.1167/iovs.15-16708. PMID 26322834
- [Derived] Tejerina AN, Vujosevic S, Varano M, Egan C, Sivaprasad S, Menon G, Massin P, Verbraak FD, Lund-Andersen H, Martinez JP, Jurgens I, Smets E, Coriat C, Wiedemann P, Agoas V, Querques G, Holz FG, Nunes S, Alves D, Neves C, Santos T, Ribeiro L, Bandello F, Cunha-Vaz J; for EVICR.net. One-year progression of diabetic subclinical macular edema in eyes with mild nonproliferative diabetic retinopathy: location of the increase in retinal thickness. Ophthalmic Res. 2015;54(3):118-23. doi: 10.1159/000438793. Epub 2015 Aug 21. PMID 26315560
- [Derived] Bandello F, Tejerina AN, Vujosevic S, Varano M, Egan C, Sivaprasad S, Menon G, Massin P, Verbraak FD, Lund-Andersen H, Martinez JP, Jurgens I, Smets RM, Coriat C, Wiedemann P, Agoas V, Querques G, Holz FG, Nunes S, Alves D, Neves C, Santos T, Ribeiro L, Cunha-Vaz J; EVICR.net. Retinal layer location of increased retinal thickness in eyes with subclinical and clinical macular edema in diabetes type 2. Ophthalmic Res. 2015;54(3):112-7. doi: 10.1159/000438792. Epub 2015 Aug 21. PMID 26315448